CLINICAL TRIAL: NCT00587379
Title: The Effect of Chronic Statin Therapy on Peripheral Arterial Tone Response to Sildenafil Citrate (Viagra), and on Erectile Function in Men With Coronary Artery Endothelial Cell Dysfunction
Brief Title: Effect of Chronic Statin and Viagra Therapy in Persons With Endothelial Cell Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed per the request of PI due to lack of participant accrual
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Amir Lerman, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 328-04; 2003-0359 - Pfizer
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Endothelial Dysfunction
Keywords: testing for Endothelial Dysfunction and coronary angiography
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients randomized to take 1 40mg Atorvastain pill per day for 6 week study period
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Patients randomized to 1 40mg placebo pill per day for 6 week study
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atorvastatin — 40 mg atorvastatin pill daily
  Arms: 1
Drug: placebo — 40 mg pill per day
  Arms: 2

SUMMARY:
To determine if 6 weeks of daily treatment with Atorvastatin 40 mg alters the immediate effect of Sildenafil Citrate (Viagra, Pfizer Inc, New York, NY) on endothelial function (activity of the artery) as measured by noninvasive peripheral arterial tonography in men and women. Also, to determine if 6 weeks of daily treatment with Atorvastatin 40 mg affects erectile function in men

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography
* No previous statin use
* Age > 18 years old
* No PDE5-1 use in the past 6 months

Exclusion Criteria:

* Patients with an Acute Coronary Syndrome
* Patients with Cardiogenic shock
* Patients > 30% coronary stenosis
* Patients with unexplained muscle pain
* Patients with acute liver disease
* Patients receiving immunosuppressant therapy, azoles, macrolide antibiotics, niacin, L-arginine
* Patients with serum creatinine > 2.0
* Patients with total cholesterol > 200 mmol/l
* Patients on current statin therapy or clinically indicated to be on statin therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
To determine if endothelial function as measured by Peripheral Arterial Tonometry improves over a 6 week period while on Atorvastatin. | 6 weeks

SECONDARY OUTCOMES:
To determine if treatment with Atovastatin affects erectile function in men | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic